CLINICAL TRIAL: NCT05829499
Title: Interventional, Non-comparative, Single-center PMCF Study to Evaluate Performance and Safety of "Xanoftal Next" Used to Attenuate Symptoms of Seasonal Allergic Conjunctivitis, Even When Associated With Dry Eye Syndrome
Brief Title: PMCF Study to Evaluate Performance and Safety of "Xanoftal Next"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C.O.C. Farmaceutici S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COC-R9-HPMC-HA
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Allergic Conjunctivitis; Dry Eye; Dry Eye Disease
MeSH Terms: conditions — Conjunctivitis, Allergic; Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eyedrops treatment arm (Experimental)
  Interventions: Device: HPMC-HA eyedrops

INTERVENTIONS:
Device: HPMC-HA eyedrops — Ocular drops based upon HPMC and HA

SUMMARY:
Dry eye disease (DED), also called keratoconjunctivitis sicca, is a multifactorial disease of the ocular surface characterized by loss of homeostasis of the tear film and accompanied by symptoms such as ocular discomfort and visual disturbance. Patients with moderate-to-severe DED may experience a reduced quality of life due to ocular pain, difficulty in performing daily activities, and depression.

Traditionally, dry eye syndrome and allergic conjunctivitis are regarded as 2 different diseases. However, recent literature has shown both conditions share similar characteristics, including several of their signs and symptoms (e.g. red, itchy, watery, and burning eyes).

On the other hand, red swollen eyelids, burning sensations, ocular irritation, loss of eyelashes and misdirected eyelashes are also common symptoms of Blepharitis, an inflammatory disorder of eyelids affecting all the age and ethnic groups.

First-line therapy for treating dry eye symptoms consists of over the counter (OTC) artificial tear drops, gels, ointments, or lubricants. Manufacturers have developed OTC products that appear to mimic the different layers of the tear film in order to maintain ocular hydration.

For these reasons, an interventional, non-comparative, Post Marketing Clinical Follow-up (PMCF) study was planned to evaluate the performance and safety of "Xanoftal Next" used to attenuate symptoms of seasonal allergic conjunctivitis, even when associated with dry eye syndrome.

The objectives of the PMCF study are confirmation of the performance, collection of additional safety data regarding expected adverse events and detection of potential unexpected adverse events associated with use of "Xanoftal Next" according to the Instructions for Use (IFU).

Each subject, after signing the Informed Consent Form, will enter the screening and baseline phase (the 2 visits will coincide) during which baseline procedures will be completed.

At baseline visit, the "Xanoftal Next" product will be administered to the enrolled subject.

The patient will perform 2 on-site visits: V0 and V2/EOS. To monitor the safety, 1 phone contact is planned (V1) to check for potential adverse events and concomitant medications intake.

ELIGIBILITY:
Inclusion Criteria:

* Signed patient Informed consent form (ICF);
* Male and Female Aged ≥ 18 years at the time of the signature of the ICF;
* Patients with ophthalmic discomfort due eye allergy or other eye discomfort caused by environmental or mechanical stress (e.g. use of computer and/or smartphone), including contact lenses wearing and blepharitis;
* Willing not to use other eye drops during the entire treatment period.

Exclusion Criteria:

* Other - different - eyes clinical conditions (e.g. glaucoma);
* Known hypersensitivity or allergy to Investigational Product (IP) components;
* Suspected alcohol or drug abuse;
* Other clinically significant and uncontrolled pathologies that may interfere with study results (e.g. rheumatic diseases, diabetes);
* Participation in another investigational study;
* Inability to follow all study procedures, including attending all site visits, tests and examinations;
* Mental incapacity that precludes adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Change in Schirmer I test: to evaluate the performance of "Xanoftal Next" to attenuate symptoms of seasonal allergic conjunctivitis, even when associated with dry eye syndrome, through the Schirmer I test | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)

SECONDARY OUTCOMES:
Change in Tear Break-up Time (TBUT): to evaluate the performance of the "Xanoftal Next" to ensure relief from ophthalmic stress, through the TBUT test | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)
Change in Ocular Surface Disease Index (OSDI): to evaluate the performance of the "Xanoftal Next" to reduce dry eye symptoms, mild to moderate, accompanied by itching, burning, foreign body sensation, redness due intrinsic or extrinsic causes | From baseline (V0 = Day 0) to 1 month (EOS/V2 = Day 30 ± 2)
  Ocular Surface Disease Index Minimum value: 0 - none of the time Maximum value: 4 - all of the time Higher scores mean a worse outcome
To evaluate the safety and tolerability of the "Xanoftal Next" through Visual Analogue Scale (VAS) - evaluation of symptoms related to dry eye disease (burning, fatigue, discomfort, redness) | End of study visit (EOS/V2 = Day 30 ± 2)
  Visual Analogue Scale Minimum value: 0 Maximum value: 10 Higher scores mean a better outcome
To evaluate the patient satisfaction through a Rensis Likert 5 points patient satisfaction scale | End of study visit (EOS/V2 = Day 30 ± 2)
  Rensis Likert 5 points patient satisfaction scale Minimum value: Very dissatisfied Maximum value: Very satisfied Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliera Policlinico Mater Domini - Università Magna Grecia di Catanzaro, Catanzaro, CZ, Italy